CLINICAL TRIAL: NCT02242747
Title: Evaluation of the Tolerability and Safety of 0.015% Ingenol Mebutate Gel Compared to 5% 5-fluorouracil Cream for the Treatment of Facial Actinic Keratosis: a Prospective Randomized Trial
Brief Title: Safety and Tolerability Study of Ingenol Mebutate Compared to 5-FU to Treat Facial Actinic Keratosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Principal Investigator, Luis Antonio Torezan, Associate Professor University of Sao Paulo, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11334
Record Dates: First submitted 2014-09-12; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis; field cancerization; ingenol mebutate; 5-fluorouracil; tolerability; safety
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ingenol mebutate (Other): Patients assigned to ingenol mebutate gel received an application a day for three consecutive days in a pre-determined area
  Interventions: Drug: ingenol mebutate
- 5% 5-FU (Other): Patients assigned to 5% 5-FU received two applications a day for four weeks in a pre-determined area
  Interventions: Drug: 5% 5-FU

INTERVENTIONS:
Drug: ingenol mebutate — an application a day for three consecutive days in a pre-determined area
  Other Names: Picato
  Arms: ingenol mebutate
Drug: 5% 5-FU — two applications a day for four weeks in a pre-determined area
  Other Names: efurix; efudex
  Arms: 5% 5-FU

SUMMARY:
Background: 5% 5-fluorouracil cream (5-FU) is a well-established treatment for actinic keratosis (AK) and ingenol mebutate gel (IMB) is a new topical field therapy.

Objective: To compare tolerability and safety of IMB with 5-FU for the treatment of facial AKs.

Methods: Open-label, prospective, randomized, controlled clinical trial with 100 patients with AKs within 25-cm2 contiguous field on the face. IMB was applied daily for three consecutive days. 5-FU was applied twice a day for four weeks. Treatment effect was evaluated at baseline and on days 2, 3, 4, 8, 15, 22, 29, 36 and 43, considering ITT populations.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 18 years
* the presence of four to eight clinically typical, visible, and discrete AKs within 25-cm2 contiguous field on the face (cheek or forehead region)
* Women with childbearing potential had to be using effective birth control and have a confirmed negative urine pregnancy test prior to trial treatment.

Exclusion Criteria:

* target treatment area was within 5 cm of an incompletely healed wound or within 10 cm of a suspected basal-cell or squamous-cell carcinoma
* if they have received previous treatment with ingenol mebutate gel on the face or scalp (previous treatment on trunk or extremities was acceptable)
* the selected treatment area had hyperkeratotic lesions or cutaneous horns and recalcitrant disease (lesions that had not responded to cryotherapy on two previous occasions)
* history or evidence of skin conditions that would interfere with the evaluation of the trial medication (e.g., eczema, unstable psoriasis, xeroderma pigmentosum)
* anticipated need for hospitalization or outpatient surgery during the first 15 days after the first trial medication application
* known sensitivity or allergy to any of the ingredients of ingenol mebutate gel or 5-FU
* presence of sunburn within of the target treatment area; current enrolment or participation in any other interventional clinical trial within 30 days of entry into this trial
* women breastfeeding
* recent use of medications or other treatments that could interfere with evaluation of the target area, such as topical medications (e.g. steroids, keratolytics, immunomodulators), artificial tanners, immunomodulators, cytotoxic drugs or interferon /interferon inducers, phototherapy, systemic retinoids, biologic/monoclonal antibody drugs, or other therapies for AKs within eight weeks prior to the first visit of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Area under the LSR (local skin reactions)-Time Curve (AUC 0-43 days) | Baseline and on day 43
  Primary endpoint was to compare the total local skin reaction grading scale (LSR) and the area under the curve (AUC) with respect to duration of effects, using a generalized linear model, assuming a logarithmic link function. Age, Fitzpatrick skin type and site of the treatment were considered as covariates. The scale ranged from 0 to 4 (with higher numbers indicating greater severity) for the following six local skin effects: erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration (maximum score of 24).

SECONDARY OUTCOMES:
Area Under the each component of the total LSR-Time Curve (AUC 0-43 days) | Baseline and on day 43
  A secondary endpoint was to evaluate and compare the AUC for each component of the total LSR using generalized linear models. The effect of treatment on the proportion of patients that completed the assigned treatment regimens was compared using generalized estimating equation model and logarithmic link function.

OTHER OUTCOMES:
Number of participants with side effects in each arm of the study | Baseline and on day 43
  An additional endpoint was to evaluate adverse effects related to the drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Antonio Torezan, PhD, Principal Investigator — Hospital das Clínicas of the University of São Paulo Medical School (HCFMUSP)
Locations (1):
- Hospital das Clínicas of the University of São Paulo Medical School (HCFMUSP), São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Samorano LP, Torezan LA, Sanches JA. Evaluation of the tolerability and safety of a 0.015% ingenol mebutate gel compared to 5% 5-fluorouracil cream for the treatment of facial actinic keratosis: a prospective randomized trial. J Eur Acad Dermatol Venereol. 2015 Sep;29(9):1822-7. doi: 10.1111/jdv.13063. Epub 2015 Feb 27. PMID 25727104